CLINICAL TRIAL: NCT00290524
Title: Prospective, Multicentric, Randomized Phase III Study Comparing Early Oral Alimentation to Nil Per Os Diet After Colorectal Surgery
Brief Title: Early Alimentation Following Colorectal Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QCTG-02-V5
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2006-04-07 (Estimated); Status verified 2006-04

CONDITIONS: Colorectal Neoplasms; Crohn Disease
Keywords: Oral alimentation following colorectal surgery; anastomosis; laparoscopy; hospitalization stay
MeSH Terms: conditions — Colorectal Neoplasms; Crohn Disease

INTERVENTIONS:
Behavioral: Oral alimentation started 12 hours after colorectal surgery

SUMMARY:
This study wants to address the question of whether or not oral alimentation should be begun early in patients following colorectal surgery compared to the classical diet which depends on reappearance of functional intestinal transit. Early oral alimentation following colorectal surgery may decrease hospitalisation stay duration.

DETAILED DESCRIPTION:
Following intestinal surgery, the classical protocol indicates the use of a naso-gastric tube and starvation more or less prolonged of the patient dependent of surgeon's view. Decision to feed the patient is based on gas and feces reappearance after surgery. However, prolonged starvation might be uncomfortable for the patient as well as increasing his hospitalization stay. Moreover, delayed feeding effect on anastomosis and wound healing is controversial and naso-gastric tube use is known to be uncomfortable and may generate secondary adverse events.

Some studies in opened surgery observed that early alimentation was beneficial against post-surgery mortality, infection risk and anastomosis dehiscence. In addition, early feeding seemed to decrease patient hospitalisation stay.

In order to conduct this study, patients having a colorectal surgery will be randomly attributed to the nil per os group, which is based on the reappearance of a functional intestinal transit, or to the experimental group, which will begin alimentation 12 hours after colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years old or more
* Class ASA (American Society of AnaesthesioIogy) I, II or III, +/- E
* Patient willing to participate in the study
* Patient who understands and accepts to sign the informed consent form
* Patient who will undergo elective or urgent colic resection using laparoscopy or opened surgery defined in section B

Section B: patient must meet one of the following inclusion criterion:

* segmental or total colorectal resection with creation of a primary colo-colic or colo-rectal anastomosis not protected with a derivation ostomy
* ileal resection in continuity with total or a segment of the colon with creation of a primary colo-colic or colo-rectal anastomosis not protected with a derivation ostomy
* Closing of a terminal or loop colostomy

Exclusion Criteria:

* Class ASA IV or V patient
* Documented problem of gastro-intestinal motility
* Pregnancy
* Any acute or recent (<10 days) septic event
* Chemotherapy during the 4 weeks preceding surgery
* Previous irradiation surrounding the planned anastomosis location
* Small intestine iatrogenic transparietal laceration done during surgery
* Small intestine synchrone resection without continuity with the colon
* Intra-peritoneal chemotherapy administered during or following surgery
* Presence of residual peritoneal carcinosis at the end of surgery
* Colic surgery associated with another major intra-abdominal surgery
* Creation of a colo-anal or ileo-anal anastomosis
* Any per-surgery discovery which requires the use of a gastric drainage procedure following surgery
* Any post-surgery change in patient condition which requires naso-gastric tube holding after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2006-01

PRIMARY OUTCOMES:
Hospitalisation stay measured in days

SECONDARY OUTCOMES:
Gastro-intestinal signs and symptoms
Treatment of gastro-intestinal signs and symptoms
Post-surgery complications

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Dubé, MD, Study Chair — Maisonneuve-Rosemont Hospital
Locations (4):
- Canada (4):
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - St-Luc Hospital, Montreal, Quebec
  - St-Sacrement Hospital, Québec, Quebec
  - Ste-Marie Hospital, Trois-Rivières, Quebec

REFERENCES:
- [Background] Habib AS, Gan TJ. Evidence-based management of postoperative nausea and vomiting: a review. Can J Anaesth. 2004 Apr;51(4):326-41. doi: 10.1007/BF03018236. PMID 15064261
- [Background] Olesen KL, Birch M, Bardram L, Burcharth F. Value of nasogastric tube after colorectal surgery. Acta Chir Scand. 1984;150(3):251-3. PMID 6464626
- [Background] Nathan BN, Pain JA. Nasogastric suction after elective abdominal surgery: a randomised study. Ann R Coll Surg Engl. 1991 Sep;73(5):291-4. PMID 1929130
- [Background] Savassi-Rocha PR, Conceicao SA, Ferreira JT, Diniz MT, Campos IC, Fernandes VA, Garavini D, Castro LP. Evaluation of the routine use of the nasogastric tube in digestive operation by a prospective controlled study. Surg Gynecol Obstet. 1992 Apr;174(4):317-20. PMID 1553612
- [Background] Petrelli NJ, Stulc JP, Rodriguez-Bigas M, Blumenson L. Nasogastric decompression following elective colorectal surgery: a prospective randomized study. Am Surg. 1993 Oct;59(10):632-5. PMID 8214960
- [Background] Pearl ML, Valea FA, Fischer M, Chalas E. A randomized controlled trial of postoperative nasogastric tube decompression in gynecologic oncology patients undergoing intra-abdominal surgery. Obstet Gynecol. 1996 Sep;88(3):399-402. doi: 10.1016/0029-7844(96)00183-4. PMID 8752247
- [Background] Cheatham ML, Chapman WC, Key SP, Sawyers JL. A meta-analysis of selective versus routine nasogastric decompression after elective laparotomy. Ann Surg. 1995 May;221(5):469-76; discussion 476-8. doi: 10.1097/00000658-199505000-00004. PMID 7748028
- [Background] Wolff BG, Pembeton JH, van Heerden JA, Beart RW Jr, Nivatvongs S, Devine RM, Dozois RR, Ilstrup DM. Elective colon and rectal surgery without nasogastric decompression. A prospective, randomized trial. Ann Surg. 1989 Jun;209(6):670-3; discussion 673-5. doi: 10.1097/00000658-198906000-00003. PMID 2658880
- [Background] Cheadle WG, Vitale GC, Mackie CR, Cuschieri A. Prophylactic postoperative nasogastric decompression. A prospective study of its requirement and the influence of cimetidine in 200 patients. Ann Surg. 1985 Sep;202(3):361-6. doi: 10.1097/00000658-198509000-00014. PMID 4037908
- [Background] Bauer JJ, Gelernt IM, Salky BA, Kreel I. Is routine postoperative nasogastric decompression really necessary? Ann Surg. 1985 Feb;201(2):233-6. doi: 10.1097/00000658-198502000-00017. PMID 3970606
- [Background] Holte K, Kehlet H. Postoperative ileus: a preventable event. Br J Surg. 2000 Nov;87(11):1480-93. doi: 10.1046/j.1365-2168.2000.01595.x. PMID 11091234
- [Background] Lacy AM, Garcia-Valdecasas JC, Pique JM, Delgado S, Campo E, Bordas JM, Taura P, Grande L, Fuster J, Pacheco JL, et al. Short-term outcome analysis of a randomized study comparing laparoscopic vs open colectomy for colon cancer. Surg Endosc. 1995 Oct;9(10):1101-5. doi: 10.1007/BF00188996. PMID 8553212
- [Background] Schwenk W, Bohm B, Haase O, Junghans T, Muller JM. Laparoscopic versus conventional colorectal resection: a prospective randomised study of postoperative ileus and early postoperative feeding. Langenbecks Arch Surg. 1998 Mar;383(1):49-55. doi: 10.1007/s004230050091. PMID 9627171
- [Background] Milsom JW, Bohm B, Hammerhofer KA, Fazio V, Steiger E, Elson P. A prospective, randomized trial comparing laparoscopic versus conventional techniques in colorectal cancer surgery: a preliminary report. J Am Coll Surg. 1998 Jul;187(1):46-54; discussion 54-5. doi: 10.1016/s1072-7515(98)00132-x. PMID 9660024
- [Background] Wexner SD, Cohen SM, Johansen OB, Nogueras JJ, Jagelman DG. Laparoscopic colorectal surgery: a prospective assessment and current perspective. Br J Surg. 1993 Dec;80(12):1602-5. doi: 10.1002/bjs.1800801238. PMID 8298938
- [Background] Moss G. Maintenance of gastrointestinal function after bowel surgery and immediate enteral full nutrition. II. Clinical experience, with objective demonstration of intestinal absorption and motility. JPEN J Parenter Enteral Nutr. 1981 May-Jun;5(3):215-20. doi: 10.1177/0148607181005003215. No abstract available. PMID 6788969
- [Background] Moore EE, Jones TN. Benefits of immediate jejunostomy feeding after major abdominal trauma--a prospective, randomized study. J Trauma. 1986 Oct;26(10):874-81. doi: 10.1097/00005373-198610000-00003. PMID 3095557
- [Background] Lewis SJ, Egger M, Sylvester PA, Thomas S. Early enteral feeding versus "nil by mouth" after gastrointestinal surgery: systematic review and meta-analysis of controlled trials. BMJ. 2001 Oct 6;323(7316):773-6. doi: 10.1136/bmj.323.7316.773. PMID 11588077
- [Background] Behrns KE, Kircher AP, Galanko JA, Brownstein MR, Koruda MJ. Prospective randomized trial of early initiation and hospital discharge on a liquid diet following elective intestinal surgery. J Gastrointest Surg. 2000 Mar-Apr;4(2):217-21. doi: 10.1016/s1091-255x(00)80059-1. PMID 10675246
- [Background] DiFronzo LA, Yamin N, Patel K, O'Connell TX. Benefits of early feeding and early hospital discharge in elderly patients undergoing open colon resection. J Am Coll Surg. 2003 Nov;197(5):747-52. doi: 10.1016/S1072-7515(03)00794-4. PMID 14585408
- [Background] Schilder JM, Hurteau JA, Look KY, Moore DH, Raff G, Stehman FB, Sutton GP. A prospective controlled trial of early postoperative oral intake following major abdominal gynecologic surgery. Gynecol Oncol. 1997 Dec;67(3):235-40. doi: 10.1006/gyno.1997.4860. PMID 9441769
- [Background] Moss G, Greenstein A, Levy S, Bierenbaum A. Maintenance of GI function after bowel surgery and immediate enteral full nutrition. I. Doubling of canine colorectal anastomotic bursting pressure and intestinal wound mature collagen content. JPEN J Parenter Enteral Nutr. 1980 Nov-Dec;4(6):535-8. doi: 10.1177/0148607180004006535. PMID 6780704
- [Background] Kiyama T, Onda M, Tokunaga A, Yoshiyuki T, Barbul A. Effect of early postoperative feeding on the healing of colonic anastomoses in the presence of intra-abdominal sepsis in rats. Dis Colon Rectum. 2000 Oct;43(10 Suppl):S54-8. doi: 10.1007/BF02237227. PMID 11052479
- [Background] Khalili TM, Navarro RA, Middleton Y, Margulies DR. Early postoperative enteral feeding increases anastomotic strength in a peritonitis model. Am J Surg. 2001 Dec;182(6):621-4. doi: 10.1016/s0002-9610(01)00818-2. PMID 11839327
- [Background] Sigalet DL, Mackenzie SL, Hameed SM. Enteral nutrition and mucosal immunity: implications for feeding strategies in surgery and trauma. Can J Surg. 2004 Apr;47(2):109-16. PMID 15132464
- [Background] Hall JC, Heel K, McCauley R. Glutamine. Br J Surg. 1996 Mar;83(3):305-12. doi: 10.1002/bjs.1800830306. PMID 8665180
- [Background] Gan TJ, Meyer T, Apfel CC, Chung F, Davis PJ, Eubanks S, Kovac A, Philip BK, Sessler DI, Temo J, Tramer MR, Watcha M; Department of Anesthesiology, Duke University Medical Center. Consensus guidelines for managing postoperative nausea and vomiting. Anesth Analg. 2003 Jul;97(1):62-71, table of contents. doi: 10.1213/01.ane.0000068580.00245.95. PMID 12818945
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2004 Jun;100(6):1573-81. doi: 10.1097/00000542-200406000-00033. No abstract available. PMID 15166580
- [Background] Kranke P, Morin AM, Roewer N, Eberhart LH. Dimenhydrinate for prophylaxis of postoperative nausea and vomiting: a meta-analysis of randomized controlled trials. Acta Anaesthesiol Scand. 2002 Mar;46(3):238-44. doi: 10.1034/j.1399-6576.2002.t01-1-460303.x. PMID 11939912
- [Background] Wildhaber BE, Yang H, Spencer AU, Drongowski RA, Teitelbaum DH. Lack of enteral nutrition--effects on the intestinal immune system. J Surg Res. 2005 Jan;123(1):8-16. doi: 10.1016/j.jss.2004.06.015. PMID 15652945
- [Background] Buck M, Houglum K, Chojkier M. Tumor necrosis factor-alpha inhibits collagen alpha1(I) gene expression and wound healing in a murine model of cachexia. Am J Pathol. 1996 Jul;149(1):195-204. PMID 8686743